CLINICAL TRIAL: NCT05382988
Title: Effect of Sodium Zirconium Cyclosilicate on Hyperkalemia After Parathyroidectomy in Secondary Hyperparathyroidism Patients With Maintenance Hemodialysis
Brief Title: Sodium Zirconium Cyclosilicate Lowers Hyperkalemia After Parathyroidectomy
Acronym: SZC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZC AFTER PTX
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Sodium Zirconium Cyclosilicate; Hyperkalemia; Hyperparathyroidism, Secondary
MeSH Terms: conditions — Hyperkalemia; Hyperparathyroidism, Secondary | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: All patients had dialysis within 24h before PTX, then were treated with PTX in Otolaryngology Head and Neck Surgery department in Guangdong Provincial People's Hospital by one experienced surgeon. The experimental group was required to take SZC 10g immediately after the blood test at 6 am, while no medical treatment was performed on patients in the control group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group was required to take SZC 10g at 6 am on the day of surgery.
  Interventions: Drug: Sodium zirconium cyclosilicate
- Control Group (No Intervention): No additional intervention was performed

INTERVENTIONS:
Drug: Sodium zirconium cyclosilicate — The experimental group was required to take SZC 10g at 6 am on the day of surgery.
  Arms: Experimental Group

SUMMARY:
Sodium zirconium cyclosilicate (SZC) has been demonstrated for its serum potassium-lowering efficacy and safety in hyperkalemia hemodialysis patients.

However, the effects of SZC during the perioperative period remained unknown.

This experiment aimed to determine whether using SZC would impact the serum potassium levels in patients with maintenance hemodialysis after parathyroidectomy (PTX).

DETAILED DESCRIPTION:
Secondary Hyperparathyroidism (SHPT) is a common and severe manifestation of chronic kidney disease (CKD), especially in end-stage renal disease (ESRD) patients. SHPT is characterized by elevated parathyroid hormone (PTH) synthesis and secretion accompanied by parathyroid cell hyperplasia.Elevated PTH level is considered as a risk factor for fracture, hyperphosphatemia, anemia, and cardiovascular calcification that worsens the health-related quality of life and increases mortality.

Parathyroidectomy (PTX) has been considered the first-line treatment for severe SHPT. Generally, approximately 29% of patients with end-stage renal disease undergo parathyroidectomy to control secondary hyperparathyroidism. Successful PTX may rapidly reduce serum PTH levels and alleviate clinical symptoms.

Postoperative hyperkalemia is one common complication after PTX. With an incidence of 25-80%, in previous research, hyperkalemia has been reported during and immediately after PTX, leading to devastating consequences.

SZC increases fecal potassium excretion and lowers serum potassium levels by binding potassium ions, demonstrated to reduce serum potassium to normal levels within 48 hours in hyperkalemia patients.

Nevertheless, the effects of SZC during the perioperative period remained unknown.

Sixty-two patients with secondary hyperparathyroidism (SHPT) were randomly recruited into the experimental and control groups. Patients in the experimental group were required to take SZC 10g before PTX. Laboratory chemistries, including serum potassium levels, serum calcium levels and serum PTH were obtained before and after surgery. We aimed to determine whether using SZC would impact the serum potassium levels in patients with maintenance hemodialysis after parathyroidectomy (PTX).

ELIGIBILITY:
Inclusion Criteria:

* Secondary Hyperparathyroidism (SHPT) is a common and severe manifestation of chronic kidney disease (CKD), especially in end-stage renal disease (ESRD) patients. ESRD MHD with SHPT patients were recruited into this study

Exclusion Criteria:

* Patients with severe cardiovascular disease who cannot tolerate general anesthesia surgery were not included in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Change of serum potassium levels | Serum potassium levels were checked at three time points, which were t0 (6 am on the day of surgery), t1 (immediate after surgery), and t2 (9 pm on the day of surgery), respectively.
  Laboratory chemistry measurement

SECONDARY OUTCOMES:
Change of serum calcium levels | Serum calcium levels were checked at three time points, which were t0 (6 am on the day of surgery), t1 (immediate after surgery), and t2 (9 pm on the day of surgery), respectively.
  Laboratory chemistry measurement

OTHER OUTCOMES:
Change of parathyroid hormone | Parathyroid hormone were checked 24h before surgery and on the first day after surgery
  Laboratory chemistry measurement

CONTACTS AND LOCATIONS:
Overall Officials: Shuangxin Liu, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang J, Li S, Su J, Xiao Z, Zhang S, Liu S, Ge P. Effect of sodium zirconium cyclosilicate on hyperkalemia after parathyroidectomy in secondary hyperparathyroidism patients with maintenance hemodialysis: A randomized trial. Medicine (Baltimore). 2024 Dec 27;103(52):e40917. doi: 10.1097/MD.0000000000040917. PMID 39969301